CLINICAL TRIAL: NCT06208930
Title: The Safety and Efficacy of Fecal Microbiota Transplantation in the Treatment of Digestive Diseases and Non-digestive System Diseases Associated With Gastrointestinal Symptoms in the Gastrointestinal Tract.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Dean of the hospital, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FMT-ALL
Record Dates: First submitted 2024-01-07; First posted 2024-01-17 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT group (Experimental)
  Interventions: Procedure: Fecal microbiota transplantation

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — Fecal microbiota transplantation (FMT) is a method for treating imbalances in the intestinal microbiota. Its basic principle involves extracting a portion of feces from a healthy individual that contains a diverse population of beneficial bacteria, processing it, and transplanting it into the digestive system of the recipient to restore a balanced intestinal microbiota.

SUMMARY:
The exploration of the safety and efficacy of fecal microbiota transplantation in the treatment of non-digestive system diseases associated with gastrointestinal symptoms in the gastrointestinal tract, while also investigating the impact of fecal microbiota transplantation on the intestinal system, and assessing the improvement of symptoms in other systems.Simultaneously optimizing the conditions during the FMT process, identifying the most effective treatment methods to enhance the therapeutic outcomes of FMT.

ELIGIBILITY:
Inclusion Criteria:

* Being able to tolerate a nasoenteric tube or swallow a capsule.

Exclusion Criteria:

* Intestinal barrier dysfunction. Inability to tolerate enteral nutrition.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Comparing the therapeutic efficacy of patients after FMT. | 0day, 7days, 30days, 3 months, 6months,12 months
  Through conducting relevant questionnaire surveys with patients, we can gain insights into the therapeutic efficacy of patients after undergoing FMT.
Comparing the differences in microbiota composition in samples such as feces and small intestinal fluid from patients. | 0day, 7days, 30days, 3 months, 6months,12 months
  Performing 16S rRNA sequencing, metagenomic sequencing, and metabolite analysis on the samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Le Wang, Shanghai, Shanghai Municipality, China